CLINICAL TRIAL: NCT04564781
Title: A Novel Multiplex Immunoassay for Predicting Intravesical BCG Response in Patients With Intermediate or High-risk Non-muscle Invasive Bladder Cancer
Brief Title: Predicting BCG Response
Status: Recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Nonagen Bioscience Corporation (Industry); University of California, San Francisco (Other); Kyoto University (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Charles Rosser, Professor, Cedars-Sinai Medical Center
Other Study IDs: CR2020-1113-0; R01CA198887 (NIH)
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Voided urine samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

SUMMARY:
To date, there are no diagnostics capable of predicting treatment response to intravesical BCG. Because of this severe limitation, nearly 50% of patients treated with BCG fail therapy and will a) require additional intravesical therapy or b) require cystectomy. A urine-based diagnostic that possesses the potential to accurately identify patients who will respond favorably to intravesical BCG is desperately needed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patients must have histologically proven Ta, carcinoma in situ (CIS) or T1 stage urothelial cell carcinoma of the bladder diagnosed within 90 days prior to scheduled BCG
* Patients must have had all grossly visible papillary tumors removed within 30 days prior to scheduled BCG or cystoscopy confirming no grossly visible papillary tumors within 30 days prior to scheduled BCG
* Patients with T1 disease must have cross-sectional imaging of abdomen/pelvis demonstrating no evidence of nodal involvement or metastatic disease (CT scan or MRI scan) within 90 days prior to scheduled BCG
* Patients must have intermediate or high-grade bladder cancer as defined by 2004 WHO/ISUP classification
* Patients must not have pure squamous cell carcinoma or adenocarcinoma.
* Patients' disease must not have micropapillary components.
* Patients must have no evidence of upper tract (renal pelvis or ureters) cancer confirmed by one of the following tests performed within 90 days prior to BCG: CT urogram, intravenous pyelogram, MR urogram, or retrograde pyelograms.
* No other prior non-bladder malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years. Patients with localized prostate cancer who are being followed by an active surveillance program are also eligible.
* Participants may be treated with immediate post-operative intravesical instillation of a chemotherapeutic agent
* Scheduled to undergo intravesical BCG therapy within 4 weeks of signing consent.
* Willing and able to give written informed consent (see Appendix 1)
* Willing to provide voided urine sample

Exclusion Criteria:

* Previous intravesical BCG therapy
* Patients must not be taking oral glucocorticoids at the time of registration.
* Patients must not be planning to receive concomitant biologic therapy, hormonal therapy, chemotherapy, surgery, or other cancer therapy while on study.
* Patients must not have known history of tuberculosis.
* Have incomplete TUR, i.e., visible residual disease
* Have had radical cystectomy
* Have a known active urinary tract infection or urinary retention
* Have active stone disease (renal or bladder) or renal insufficiency (creatinine >2.0 mg/dL) - Serum creatinine value can be up to 2 years before consent, otherwise repeat.
* Have ureteral stents, nephrostomy tubes or bowel interposition
* Have recent genitourinary instrumentation (within 7 days prior to signing consent)
* Be unable or unwilling to complete BCG induction and maintenance regimen

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recently diagnosed intermediate or high risk non-muscle invasive bladder cancer, who are destined to undergo intravesical BCG therapy.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-09-18 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of multiplex immunoassay will be confirmed by surveillance cystoscopy. | present through 04/30/2027

SECONDARY OUTCOMES:
Sensitivity and specificity of multiplex immunoassay will be compared to panel of urinary cytokines. | present through 04/30/2027

CONTACTS AND LOCATIONS:
Overall Officials: Charles Rosser, MD, Study Director — Nonagen Bioscience Corporation; Hideki Furuya, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (5):
- United States (4):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - UCSF, San Francisco, California
  - University of Texas Southwestern, Dallas, Texas
- Kyoto University, Kyoto, Kyoto, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Furuya H, Sakatani T, Tanaka S, Murakami K, Waldron RT, Hogrefe W, Rosser CJ. Bladder cancer risk stratification with the Oncuria 10-plex bead-based urinalysis assay using three different Luminex xMAP instrumentation platforms. J Transl Med. 2024 Jan 2;22(1):8. doi: 10.1186/s12967-023-04811-2. PMID 38167321
- [Derived] Furuya H, Sakatani T, Tanaka S, Murakami K, Waldron RT, Hogrefe W, Rosser CJ. Bladder cancer risk stratification with the Oncuria 10-plex bead-based urinalysis assay using three different Luminex xMAP instrumentation platforms. Res Sq [Preprint]. 2023 Nov 25:rs.3.rs-3635581. doi: 10.21203/rs.3.rs-3635581/v1. PMID 38045238